CLINICAL TRIAL: NCT05958615
Title: Evaluation of Feasibility, Acceptability, and Preliminary Efficacy of a Dyadic Positive Psychology Intervention for Patients Post-bariatric Surgery and Their Partners: A Pilot Randomized Controlled Trial
Brief Title: Positive Psychology Intervention for Patients Post-bariatric Surgery and Their Partners
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa McGarrity, Ph.D. (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor-Investigator, Larissa McGarrity, Ph.D., Principal Investigator, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB_00165737; 1K12TR004413 (NIH)
Record Dates: First submitted 2023-07-11; First posted 2023-07-24 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Waitlist Control Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Condition (Experimental): Participants will receive 8 weeks of ReConnect followed by 8 weeks check-in surveys/follow-ups, as well as 3 assessments (baseline, 8 weeks, 16 weeks).
  Interventions: Behavioral: Reimagining Us in the Context of Bariatric Surgery (ReConnect)
- Waitlist Control Condition (Other): Participants will receive 8 weeks of check-in surveys/follow-ups followed by 8 weeks of ReConnect, as well as 3 assessments (baseline, 8 weeks, 16 weeks).
  Interventions: Behavioral: Reimagining Us in the Context of Bariatric Surgery (ReConnect)

INTERVENTIONS:
Behavioral: Reimagining Us in the Context of Bariatric Surgery (ReConnect) — ReConnect is an intervention for bariatric surgery patients approximately 2 years after surgery and their romantic partners to participate in together with the goal of improving mental health and enhancing resilience. The intervention is entirely remotely-delivered via handouts sent by PDF and mail to participants instructing them through the 8 weekly modules, as well as associated videos. Each module features psychoeducational materials, instructions and guidance on positive psychology activities, choices of activities to complete both individually and as a couple, and additional resources relevant to that week's theme. The themes are: channeling strengths and focusing on the positive, clarifying values and finding meaning, goal setting, intimacy and fostering the relationship, open communication and gratitude, self-care and savoring the moment, fostering relationships and acts of kindness, and maintaining progress long-term.

SUMMARY:
The goal of this waitlist-control design, pilot randomized controlled trial is to test feasibility, acceptability, and preliminary efficacy of a remotely-delivered dyadic positive psychology intervention for patients 2 years after bariatric surgery and their romantic partners (called ReConnect).

The main question it aims to answer is whether the intervention results in improvements in depressive symptoms for patients and partners. The additional questions it aims to answer are whether the intervention results in improvements in resilience, relationship satisfaction, eating and physical activity behaviors, and weight maintenance for those in the intervention versus waitlist control condition.

Participant couples randomly assigned to the intervention condition will engage in ReConnect for 8 weekly modules and associated positive psychology activities, some individually and some as a couple. Participant couples randomly assigned to the waitlist control condition will wait for 8 weeks to begin the 8 week intervention. All participants will fill out assessment measures at baseline, 8 weeks, and 16 weeks.

DETAILED DESCRIPTION:
Bariatric surgery is the most effective intervention for severe obesity and associated co-morbidities. However, around 2 years after surgery, a substantial proportion of patients struggle with weight regain, psychological complications (e.g., disordered eating, depression), and relationship challenges. To achieve optimal long-term outcomes, a biopsychosocial focus and treatment approach is critical. Existing interventions primarily target weight, occur at the individual patient level, use a risk-based or problem-focused lens, and are inaccessible to the average patient. In contrast, this proposed research will test feasibility, acceptability, and preliminary efficacy of an intervention to improve psychosocial health, occurring at the dyadic (patient and partner) level, using a strengths-based or positive psychology lens, and remotely-delivered for accessibility. This multi-faceted approach is needed to address the high rate of psychiatric disorders and lack of social support among bariatric surgery patients that compromises long-term surgical outcomes. Patients in relationships report inconsistency in support provision from partners, lose less weight than those not in relationships, and are at elevated risk of divorce post-surgery. The investigator(s) research has demonstrated declines in relationship satisfaction from before to after surgery, and associations with elevated levels of binge eating, anxiety, and social stress 2 years after surgery. The investigator(s) has also documented the importance of adaptive coping, social support, and resilience for improved mental health and eating behaviors in this stigmatized population. In combination, existing research supports the need for dyadic-level and strengths-focused intervention to prevent exacerbation of psychological distress and difficulties in long-term weight management.

The investigator and research team have utilized pilot grant funding to adapt an evidence-based dyadic positive psychology intervention (dPPI) for post-bariatric surgery patients and their partners. This intervention was developed in a two-phase, mixed-methods study. The investigator first obtained feedback from 6 patients and partners in focus groups about relationship health following bariatric surgery and intervention needs. The investigators then asked these couples to pilot test 4 adapted intervention modules and obtained quantitative and qualitative feedback, which suggested high satisfaction with and benefit from the intervention modules. This study resulted in a finalized 8-module, remotely-delivered dPPI with content consisting of activities (expressing gratitude, practicing acts of kindness, fostering relationships, focusing on the positive, savoring, working toward goals, meaning finding/values, planning for the future) completed individually and as a couple. The dPPI is now ready for formal testing of feasibility, acceptability, and preliminary efficacy in a pilot randomized clinical trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Adult couples (18 years and older) consisting of one partner who had bariatric surgery (Roux-en-Y gastric bypass or sleeve gastrectomy) at participating institution
* Between 1 to 3 years post bariatric surgery performed at participating institution and
* A cohabiting romantic partner who have been in the same relationship from before bariatric surgery to time of recruitment
* Both partners are willing and able to enroll in study

Exclusion Criteria:

* Couples in which both members have undergone bariatric surgery
* Current participation in another intervention study
* Lack of access to internet for remotely delivered intervention

  * Absence of depressive symptoms, relationship challenges, or difficulty coping with lifestyle changes at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptoms | Baseline
  Patient Health Questionnaire-9 (PHQ-9) Measured Scale 0 - 27 (0 = minimum - 27 maximum), the higher the score the worse outcome.
Depressive Symptoms | Week # 8
  Patient Health Questionnaire-9 (PHQ-9) Measured Scale 0 - 27 (0 = minimum - 27 maximum), the higher the score the worse outcome.
Depressive Symptoms | Week #16
  Patient Health Questionnaire-9 (PHQ-9) Measured Scale 0 - 27 (0 = minimum - 27 maximum), the higher the score the worse outcome.

SECONDARY OUTCOMES:
Resilience | Baseline
  Connor-Davidson Resilience Scale (CD-RISC) Measured Scale 0 -100 (0 = minimum - 100 = maximum), the higher the score the better outcome.
Resilience | Week # 8
  Connor-Davidson Resilience Scale (CD-RISC) Measured Scale 0 -100 (0 = minimum - 100 = maximum), the higher the score the better outcome.
Resilience | Week # 16
  Connor-Davidson Resilience Scale (CD-RISC) Measured Scale 0 -100 (0 = minimum - 100 = maximum), the higher the score the better outcome.
Relationship Satisfaction | Baseline
  Dyadic Adjustment Scale (DAS) Measured Scale 0-151 ((0 = minimum - 151 = maximum), the higher the score the better outcome.
  the minimum and maximum values, and whether higher scores mean a better or worse outcome.
Relationship Satisfaction | Week #8
  Dyadic Adjustment Scale (DAS) Measured Scale 0-151 ((0 = minimum - 151 = maximum), the higher the score the better outcome.
  the minimum and maximum values, and whether higher scores mean a better or worse outcome.
Relationship Satisfaction | Week #16
  Dyadic Adjustment Scale (DAS) Measured Scale 0-151 ((0 = minimum - 151 = maximum), the higher the score the better outcome.
  the minimum and maximum values, and whether higher scores mean a better or worse outcome.
Physical Activity | Baseline
  Leisure Time Physical Activity Questionnaire is an assessment change from initial baseline measure.
Physical Activity | Week #8
  Leisure Time Physical Activity Questionnaire is an assessment change from initial baseline measure.
Physical Activity | Week #16
  Leisure Time Physical Activity Questionnaire is an assessment change from initial baseline measure.
Eating Behaviors | Baseline
  Short Healthy Eating Index Survey Measured Scale 0 -100 (0 = minimum - 100 = maximum), the higher the score the better outcome.
Eating Behaviors | Week # 8
  Short Healthy Eating Index Survey Measured Scale 0 -100 (0 = minimum - 100 = maximum), the higher the score the better outcome.
Eating Behaviors | Week # 16
  Short Healthy Eating Index Survey Measured Scale 0 -100 (0 = minimum - 100 = maximum), the higher the score the better outcome.
Weight Maintenance | Baseline
  Percent Excess Weight Loss. Change will be assessed from initial reported weight.
Weight Maintenance | Week #8
  Percent Excess Weight Loss. Change will be assessed from initial reported weight.
Weight Maintenance | Week #16
  Percent Excess Weight Loss. Change will be assessed from initial reported weight.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa McGarrity, PhD, Principal Investigator — University of Utah Craig Neilsen H. Rehabilitation Hospital
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No